CLINICAL TRIAL: NCT03415997
Title: Dosing Iodinated Contrast Media According to Lean vs. Total Body Weight at Abdominal CT: a North American Randomized Controlled Trial
Brief Title: Dosing Iodinated Contrast Media According to Lean vs. Total Body Weight
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Andreu Costa, Principal Investigator; Section Head of Abdominal Radiology, Queen Elizabeth II Health Sciences Centre; Assistant Professor, Dalhousie University, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: NSHA REB 1023119
Record Dates: First submitted 2018-01-18; First posted 2018-01-30 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Contrast Media Dosing
MeSH Terms: interventions — Iohexol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Total Body Weight (Active Comparator)
  Interventions: Drug: Iohexol
- Lean Body Weight (Active Comparator)
  Interventions: Drug: Iohexol

INTERVENTIONS:
Drug: Iohexol — Iodinated contrast media

SUMMARY:
The purpose of this study is to evaluate the effect of dosing iodinated contrast media according to a patient's total body weight vs. lean body weight. Participants will be randomized into 2 groups based on contrast dosing technique, and solid organ enhancement at uniphasic abdominal CT will be measured.

ELIGIBILITY:
Inclusion Criteria:

* outpatients only
* patients scanned on modern Siemens scanners at our institution

Exclusion Criteria:

* self-reported history of chronic kidney, heart or liver disease
* allergy to iodinated contrast
* acute illness
* outside maximum threshold limit for weight-based contrast dosing
* pregnancy
* image degradation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 239 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Mean hepatic enhancement (MHE): difference in liver attenuation on computed tomography images acquired before and after administration of contrast (in portal venous phase), as measured in Hounsfield units (HU) | 1 hour
  Images of the liver will be obtained before and after administration of iodinated contrast media. Regions of interest will be drawn on these pre- and post- contrast computed tomography (CT) images of the liver. The average attenuation before and after contrast administration will be calculated. The mean hepatic enhancement (MHE) will be calculated as the average attenuation post-contrast minus the average attenuation pre-contrast. This will provide a measure of liver enhancement.

SECONDARY OUTCOMES:
Standard deviation in mean hepatic enhancement (sigma MHE): standard deviation in the difference in liver attenuation on CT acquired before and after administration of contrast (in portal venous phase), as measured in Hounsfield units (HU) | 1 hour
  Images of the liver will be obtained before and after administration of iodinated contrast media. Regions of interest will be drawn on these pre- and post- contrast computed tomography images of the liver. The average attenuation before and after contrast administration will be calculated. The mean hepatic enhancement (MHE) will be calculated as the average attenuation post-contrast minus the average attenuation pre-contrast. The standard deviation in MHE will provide a measure of inter-patient variability.

CONTACTS AND LOCATIONS:
Overall Officials: Andreu Costa, Md FRCPC, Principal Investigator — Nova Scotia Health Authority
Locations (1):
- Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Costa AF, Peet K, Abdolell M. Dosing Iodinated Contrast Media According to Lean Versus Total Body Weight at Abdominal CT: A Stratified Randomized Controlled Trial. Acad Radiol. 2020 Jun;27(6):833-840. doi: 10.1016/j.acra.2019.07.014. Epub 2019 Aug 19. PMID 31439467